CLINICAL TRIAL: NCT07267806
Title: Camrelizumab and Apatinib With or Without FOLFOX Chemotherapy as First-Line Treatment for Advanced Hepatocellular Carcinoma (HCC): A Randomized, Controlled, Open-Label, Multicenter Phase III.
Brief Title: Camrelizumab and Apatinib With or Without FOLFOX Chemotherapy for Advanced HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Linhui Peng (Other)
Responsible Party: Sponsor-Investigator, Linhui Peng, Associate Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-787-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Hepato Cellular Carcinoma (HCC); Chemotherapy Effect
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Intervention Model Description: Arm1: infusional FOLFOX plus Camrelizumab and Apatinib Arm2: Camrelizumab and Apatinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infusional FOLFOX (Experimental): Infusional mFOLFOX7 plus Camrelizumab and apatinib
  Interventions: Drug: Infusional mFOLFOX7 plus Camrelizumab and apatinib
- Excluding FOLFOX (Active Comparator): Camrelizumab and Apatinib
  Interventions: Drug: Camrelizumab and apatinib

INTERVENTIONS:
Drug: Infusional mFOLFOX7 plus Camrelizumab and apatinib — Oxaliplatin 85mg/m2 IV on Days 1 of a 21 day cycle Fluorouracil 5-FU continuous infusion: 400mg/m2 on Dand then 2400mg/m2 for 46h of each 21 day cycle. this chemotherapy regimen should be administered for a maximum of 6 cycles. Camrelizumab 200mg infusion on D1 forevery 21 days Apatinib 250mg, po, qd for every 21 days.
  Arms: Infusional FOLFOX
Drug: Camrelizumab and apatinib — Camrelizumab 200mg infusion on D1 forevery 21 days Apatinib 250mg, po, qd for every 21 days.
  Arms: Excluding FOLFOX

SUMMARY:
This is a multi-center randomized phase III clinical study of first-line Camrelizumab and Apatinib with or without intravenous FOLFOX Chemotherapy for Advanced Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. ≥18 years old, male and female;
3. Before treatment, it was confirmed by histopathology or cytology, or clinically diagnosed as hepatomegaly.Patients with Hepatocellular Carcinoma, HCC);
4. BCLC stage B or C hepatocellular carcinoma, which is not suitable for curative surgical or local therapies, or has progressed after such treatments.
5. Local therapy (including but not limited to surgery, radiation therapy, transarterial chemoembolization [TACE], hepatic arterial infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) must have been completed at least 4 weeks prior to the baseline radiographic scan (with the exception of palliative radiotherapy, for which a 2-week interval is sufficient)."
6. Has not received any systemic treatment for HCC.
7. According to RECIST 1.1 standard, patients have at least one measurable lesion (CT/MRI scan long diameter ≥10mm or CT/MRI scan short diameter ≥15mm for lymph node lesions, and the lesion has not received radiotherapy, freezing or other local treatments);
8. Child-pugh liver function grading: Grade A or Grade Better B (≤7 points)
9. ECOG PS score 0-2;
10. Expected survival ≥ 12 weeks;
11. Major organ functions are basically normal and meet the following requirements (within 7 days before starting the study treatment):

    1. Complete blood count: absolute neutrophil count ≥ 1.5*10^9/L, platelets (PLT) ≥ 75*10^9/L, hemoglobin ≥ 90 g/L;
    2. Blood biochemistry: albumin ≥ 25 g/L; total bilirubin ≤ 3.0 × upper limit of normal (ULN); alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 5 × ULN; creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CrCl) > 50 mL/min.
    3. International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) no more than 6 seconds above the normal control range;
    4. Urine protein <2 (if urine protein ≥2, a 24-hour urine protein quantification can be performed; 24-hour urine protein <1.0 g is allowed for inclusion).
12. Patients with active hepatitis B virus (HBV) infection must receive anti-HBV therapy prior to initiating study treatment and be willing to continue antiviral therapy throughout the study; hepatitis C virus (HCV) RNA-positive patients must receive antiviral therapy according to local standard treatment guidelines with liver function not exceeding CTCAE grade 1 elevation.
13. Women of childbearing potential should have a negative serum or urine pregnancy test within 7 days prior to study enrollment, must not be breastfeeding, and must agree to use contraception during the study and for 6 months after the study; men must agree to use contraception during the study and for 6 months after the study.

    -

Exclusion Criteria:

1. Known cholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma, and fibrolamellar carcinoma; having other active malignancies within the past 5 years or simultaneously, excluding HCC. Successfully treated localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc., can be included.
2. Patients who are preparing for or have previously undergone organ or allogeneic hematopoietic stem cell transplantation;
3. Patients with clinical symptoms of moderate to severe ascites that require therapeutic puncture or drainage; uncontrolled pleural effusion or pericardial effusion of moderate amount or more;
4. Patients with a history of gastrointestinal bleeding within 6 months before the start of the study treatment or a clear tendency for gastrointestinal bleeding, such as: high-risk or severe esophageal and gastric varices, localized active gastrointestinal ulcer lesions, or persistent positive fecal occult blood;
5. Patients who have had abdominal fistulas, gastrointestinal perforation, or intra-abdominal abscesses within 6 months before the start of the study treatment;
6. Patients with known hereditary or acquired bleeding disorders (such as coagulation dysfunction) or thrombophilia.
7. Currently using or having recently used (within 10 days before the start of the study treatment) aspirin [>325 mg/day (maximum antiplatelet dose)] or dipyridamole, ticlopidine, clopidogrel, and cilostazol;
8. Occurrence of thrombotic or embolic events within 6 months before the start of the study treatment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction, pulmonary .embolism).
9. Uncontrolled cardiac clinical symptoms or conditions, such as:

   1. Heart failure of NYHA class II or above;
   2. Unstable angina;
   3. Myocardial infarction occurring within the past year;
   4. Clinically significant supraventricular or ventricular arrhythmias requiring medical intervention;
   5. Patients with hypertension whose condition is poorly controlled by medication and who are assessed by a doctor to be at high risk when using apatinib;
10. Suffering from hypertension that cannot be well controlled with antihypertensive medication (systolic ≥140 mmHg or diastolic ≥90 mmHg); history of hypertensive crises or hypertensive encephalopathy;
11. Major vascular disease occurring within 6 months prior to the start of study treatment (e.g., an aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis);
12. Severe, non-healing, or dehisced wounds, as well as active ulcers or untreated fractures;
13. Undergoing major surgery (except for diagnosis) within 4 weeks before the start of study treatment or anticipated need for major surgery during the study period;
14. Inability to swallow pills, malabsorption syndrome, or any condition affecting gastrointestinal absorption;
15. History of intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months before starting study treatment;
16. Evidence of intra-abdominal gas that cannot be explained by puncture or recent surgery;
17. Past or present central nervous system metastases; 18. History of hepatic encephalopathy.
18. Currently accompanied by interstitial pneumonia or interstitial lung disease, or with a history of interstitial pneumonia or interstitial lung disease requiring steroid treatment, or other conditions that may interfere with the assessment and management of immune-related lung toxicity, such as pulmonary fibrosis, organizing pneumonia, pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or severely impaired lung function; active tuberculosis;
19. Currently accompanied by interstitial pneumonia or interstitial lung disease, or with a history of interstitial pneumonia or interstitial lung disease requiring steroid treatment, or other conditions that may interfere with the assessment and management of immune-related lung toxicity, such as pulmonary fibrosis, organizing pneumonia, pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or severely impaired lung function; active tuberculosis;
20. Subjects with active autoimmune diseases or a history of autoimmune diseases that may relapse (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects whose condition can be controlled solely with hormone replacement therapy may be included]); subjects with skin diseases that do not require systemic treatment such as vitiligo, psoriasis, or alopecia, subjects with type 1 diabetes controlled with insulin therapy, or subjects whose childhood asthma has fully resolved and require no intervention as adults may be included; subjects with asthma requiring medical intervention with bronchodilators cannot be included.
21. Use of immunosuppressants or systemic steroid therapy within 14 days prior to the start of study treatment to achieve immunosuppression (dose >10 mg/day of prednisone or other equivalent steroids);
22. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications; oral or intravenous therapeutic antibiotics within 2 weeks prior to the start of study treatment (patients receiving prophylactic antibiotics are eligible for the study, such as for prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease);
23. Congenital or acquired immunodeficiency (e.g., HIV infection);
24. Coinfection with hepatitis B and hepatitis C;
25. Prior treatment with other anti-PD-1 antibodies or other PD-1/PD-L1 targeted immunotherapies, or prior treatment with apatinib;
26. Vaccination with live attenuated vaccines within 28 days prior to the start of study treatment, or anticipated need for such vaccines during camrelizumab treatment or within 60 days after the last dose of camrelizumab;
27. Treatment with other investigational drugs within 28 days prior to the start of study treatment.
28. According to the researcher's judgment, the patient has other factors that may affect the study results or lead to premature termination of the study, such as alcoholism, drug abuse, other severe illnesses (including psychiatric disorders) requiring combined treatment, significant abnormalities in laboratory tests, or family or social factors that could affect the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 3 years
  The time from the start of treatment to the first progression of the patient's diseaseTime based on RECIST V1.1.
Overall Survival(OS) | up to approximately 5 years
  The time between the start of treatment and the patient's deathTime.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | up to approximately 3 years
  ORR is defined as the proportion of patients who achieve a reduction in tumor size by a predefined amount within the shortest time frame based on REClSTv1.1. ORR is defined as the sum of partial response (PR) and complete response (CR), that is, the proportion of patients who achieve either PR or CR.
During of response(DOR) | up to approximately 3 years
  how long a disease continues to respond to a treatment after the initial response is achieved, without the disease getting worse again based on RECIST v1.1.
Disease control rate(DCR) | up to approximately 3 years
  The percentage of patients whose tumors shrink or stabilize for a certain period otime, including complete response (CR), partial response (PR), and stable (SD) cases. Patientswere evaluated once every 3 cycles during the 1st to 6th treatment cycle and once every 3months during the sequential treatment phase.
Time to progression(TTP) | up to approximately 3 years.
  It is defined as the time from the start of treatment (or randomisation) until the objective documentation of disease progression based on RECIST v1.1.
Progression-Free Survival based on mRECIST(mPFS) | up to approximately 3 years
  The time from the start of treatment to the first progression of the patient's diseaseTime based on mRECIST
Time to progression based on mRECIST(mTTP) | up to approximately 3 years.
  It is defined as the time from the start of treatment (or randomisation) until the objective documentation of disease progression based on mRECIST.
Disease control rate based on mRECIST(mDCR) | up to approximately 3 years
  The percentage of patients whose tumors shrink or stabilize for a certain period otime, including complete response (CR), partial response (PR), and stable (SD) cases based on mRECIST. Patientswere evaluated once every 3 cycles during the 1st to 6th treatment cycle and once every 3months during the sequential treatment phase.Time Frame: up to approximately 3 years
During of response based on mRECIST(mDOR) | up to approximately 3 years
  how long a disease continues to respond to a treatment after the initial response is achieved, without the disease getting worse again based on mRECIST .
Objective Response Rate based on mREClST(mORR) | up to approximately 3 years
  ORR is defined as the proportion of patients who achieve a reduction in tumor size by a predefined amount within the shortest time frame based on mREClST. ORR is defined as the sum of partial response (PR) and complete response (CR), that is, the proportion of patients who achieve either PR or CR.
6 months Progression-Free Survival Rate(6-mon-PFSR) | up to approximately 3 years
  The incidence of disease progression within the first 6 months of the patient's treatment.
12 months Progression-Free Survival Rate(12-mon-PFSR) | up to approximately 3 years
  The incidence of disease progression within the first 12 months of the patient's treatment.
18 months Progression-Free Survival Rate(18-mon-PFSR) | up to approximately 3 years.
  The incidence of disease progression within the first 18 months of the patient's treatment.
12 months Overall Survival Rate(12-mon-OSR) | 2 years
  Proportion of patients surviving from the start of enrollment to the full 12 months of follow-up.
24 months Overall Survival Rate(24-mon-OSR) | 2 years.
  Proportion of patients surviving from the start of enrollment to the full 24 months of follow-up.
36 months Overall Survival Rate(36-mon-OSR) | 3 years.
  Proportion of patients surviving from the start of enrollment to the full 36 months of follow-up.
Treatment-related Adverse Event(TRAE) | up to approximately 3 years.
  The classification of adverse events during treatment was based on NCI-CTCAE v5.0 criteria.
Surgical Conversion Rate | up to approximately 3 years.
  Conversion of initially unresectable patients to resection.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No